CLINICAL TRIAL: NCT01004484
Title: Physiological Effects of Yogurt Containing Bifidobacterium Lactis (Bb12) in Subjects With Non-Diarrhea Functional Gastrointestinal Symptoms
Brief Title: Physiological Effects of Yogurt With Bb12 in Subjects With GI Symptoms Strointestinal Symptoms
Acronym: GM-WGTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: General Mills (Industry)
Responsible Party: Tamar Ringel-Kulka, MD, MPH, The University of North Carolina at Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 09-0480
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Non-diarrhea Functional Bowel Symptoms
Keywords: non-patients; non-diarrhea functional bowel symptoms
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yogurt with probiotics and inulin (Active Comparator): A probiotic yogurt containing Streptococcus thermophilus and Lactobacillus bulgaricus (at least 1x10^8 cfu/g); the probiotic bacteria Bifidobacterium lactis (Bb12) (5x10^7 cfu/g; 5x10^9 cfu/serving) and Inulin (3gr/serving).
  Interventions: Other: A probiotic yogurt with inulin
- Placebo (Placebo Comparator): Acidified dairy snack without yogurt cultures, probiotic or inulin.
  Interventions: Other: Acidified dairy snack

INTERVENTIONS:
Other: A probiotic yogurt with inulin — A 4 oz. cup with a probiotic yogurt containing Streptococcus thermophilus and Lactobacillus bulgaricus (at least 1x10^8 cfu/g); the probiotic bacteria Bifidobacterium lactis (Bb12) (5x10^7 cfu/g; 5x10^9 cfu/serving) and Inulin (3gr/serving), once daily.
  Arms: Yogurt with probiotics and inulin
Other: Acidified dairy snack — A 4 oz. cup of acidified dairy snack, once daily.
  Arms: Placebo

SUMMARY:
Hypothesis:

* Daily consumption of yogurt containing probiotic bacteria (Bb12) and inulin will significantly decrease whole gut and intestinal segmental transit time
* The effect of accelerating intestinal transit will be associated with other GI physiology parameters including stool frequency and stool consistency.

DETAILED DESCRIPTION:
In previous preliminary study we have shown that daily consumption of a probiotic yogurt drink containing probiotic bacteria (Bifidobacterium lactis Bb12) and inulin significantly accelerate colonic transit time in non-patients population with functional bowel symptoms. In this study we investigate the physiologic effect(s) of yogurt with the same bacteria and inulin on gastrointestinal function by assessing its effect on the whole gut and segmental transit time using SmartPill™ - a recently introduced device of measuring intestinal transit time. The proposed study will provide additional information on the effect on the whole gut transit as well as on other segments of the GI tract (stomach and small bowel). Assessment of transit time in the proposed study will be done following 10 to 14 days of the probiotic yogurt consumption.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. 18 - 70 y/o.
3. Existing functional GI symptoms for at least two weeks.
4. No current prescription treatment of functional GI Symptoms. Over the counter (OTC) medications allowed if still symptomatic despite current OTC therapy.
5. Normal colonoscopy within the last 3 years if age >50.
6. Normal initial screening evaluation including medical history, physical examination, and laboratory tests (CBC, ESR, blood chemistry including BUN, electrolytes, serum creatinine, bilirubin, ALT, AST, ALP, amylase, lipase, TSH, and routine stool microbiology).

Exclusion Criteria:

1. Physician treatment of functional bowel symptoms in the last 10 months.
2. Current use of prescription medications for functional bowel symptoms.
3. 1 or more bowel movements per day.
4. Contraindication to use of Fleets Enema or the balloon expulsion test.
5. Severe difficulty with defecation and/or recurrent events of unsuccessful defecation with straining.
6. Severe FBD symptoms at baseline.
7. Medical diagnosis of FBD
8. Daily use of OTC anti-pain, anti-diarrheal or laxative medications.
9. Presence of pre-existing serious, unstable medical condition.
10. Insulin-dependent Diabetes Mellitus.
11. Current diagnosis of major psychiatric disorder or suicide attempt within the last two years.
12. History of alcohol or substance abuse within two years.
13. Treatment for malignancy other than BCC or SCC within the last 5 years.
14. Self-diagnosis of lactase deficiency that explains symptoms (i.e., symptoms resolved or reduced significantly with lactose-free diet.)
15. Participation in a drug study within the last 21 days.
16. Antibiotic treatment or probiotic products consumption during the last 4 weeks.
17. Predisposition to infection (i.e. immune system compromised, rheumatic heart disease, artificial valve, history of bacterial endocarditis, active bacterial disease, etc).
18. History of gastric bezoar (masses trapped in the gastrointestinal tract).
19. Disorders of swallowing and/or severe difficulty swallowing (dysphagia) food or pills.
20. Suspected strictures, fistulas, colon cancer or other physiological GI obstruction.
21. Allergies to components of the Smart Bar: Granola (Rolled Oats, Evaporated Cane Juice, Expeller Pressed Canola Oil, Defatted Wheat Germ, Oat Flour, Brown Rice Syrup, Molasses, Salt, Natural Flavor, Soy Lecithin), Whey Crisp, Rice Syrup, Corn Syrup, Whey Protein Isolate, Invert Sugar, Puffed Wheat, Apples, Maltodextrin, Sorbitol, Apple Juice Concentrate, Partially Hydrogenated Vegetable Oil (Cottonseed, Soybean), Honey, Natural and Artificial Flavor, Salt, Vanilla.
22. Prior GI surgery except for removal of gall bladder or appendix; prior stomach surgery for acid reflux disease (Nissen fundoplication).
23. Abdominal surgery within the past 3 months.
24. History of inflammatory bowel disease.
25. History of inflammation of the lining of the gastrointestinal tract (diverticulitis or diverticulosis), tightening of bowels (diverticular stricture), and other intestinal strictures (per self report).
26. Body Mass Index (BMI) > 40
27. Female of childbearing age not practicing birth control and/or pregnant or lactating.
28. Cardiovascular, endocrine, renal, or other chronic disease likely to affect GI motility.
29. Use of medical device such as a pacemaker, infusion pump, or insulin pump.
30. Use of following prohibited medications for 1 day prior to the SmartPill ingestion and the day of SmartPill ingestion: (a) Medication to alter gastric pH (Proton Pump Inhibitors); (b) antacids;
31. Use of following prohibited medications for 3 days prior to the SmartPill ingestion and the day of SmartPill ingestion (a) Medication to lower stomach; (b) Medication that affect GI motility

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures will be the whole gut (WGTT) and colonic transit time (CTT) as assessed by SmartPill™ | 10-28 days

SECONDARY OUTCOMES:
Secondary outcome measures (a) Stool frequency (b) Stool consistency (c) Gastric emptying and small bowel transit time | 10-28 days

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Ringel-Kulka, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-CH Program of Digestive Health, Chapel Hill, North Carolina, United States